CLINICAL TRIAL: NCT01040169
Title: Clinical Efficacy of a Toothpaste on Hypersensitivity Reduction
Acronym: Yeaple
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-0308-SF-PROC-SEN-ED
Record Dates: First submitted 2008-09-27; First posted 2009-12-29 (Estimated); Results first posted 2009-12-29 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nupro C Prophylaxis paste (Placebo Comparator): Fluoride Free
  Interventions: Device: Mint Prophy paste - Fluoride free
- ProClude Prophylaxis paste (Experimental): Arginine
  Interventions: Device: Arginine/Calcium Carbonate

INTERVENTIONS:
Device: Arginine/Calcium Carbonate — One application
  Arms: ProClude Prophylaxis paste
Device: Mint Prophy paste - Fluoride free — one application
  Other Names: Nupro C Prophylaxis paste - Fluoride free
  Arms: Nupro C Prophylaxis paste

SUMMARY:
Tooth sensitivity reduction after dentifrices use

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.
* Availability for the three month duration of the study.
* Two sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to tactile stimuli (Yeaple probe) as defined by a score between 10-50gms. of force.
* Qualifying response to the air blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both the parameters assessed (tactile or air) on two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for three months prior to entry into the study.
* Signed Informed Consent Form.

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Subjects that began to take anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily analgesics within one month prior to the start of the study or who have to start taking these during the course of the study.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past three months.
* Current participation in any other clinical study.
* Pregnant or lactating subjects.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schiff, DMD, Principal Investigator
Locations (1):
- Jacobsen Dental Clinic, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment, screening and enrollment completed at the clinic site
Groups:
- Nupro C Prophylaxis Paste; ProClude Prophylaxis Paste: single, unit dose application professionally applied to the teeth (by a dentist)at the beginning of the study
Period: Overall Study
Arm/Group | Nupro C Prophylaxis Paste | ProClude Prophylaxis Paste
Started | 35 | 44
Completed | 32 | 36
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nupro C Prophylaxis Paste | ProClude Prophylaxis Paste | Total
Number analyzed (Participants) | 35 | 44 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 35 | 43 | 78.0
  >=65 years | 0 | 1 | 1.0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.34 (9.1) | 35.55 (8.9) | 36.34 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 15 | 23 | 38
Region of Enrollment [Number; unit: participants]
  United States | 35 | 44 | 79

OUTCOME MEASURES:

1. Primary Outcome: Tooth Hypersensitity to Touch Stimuli (Tactile)
Description: Units on a scale:Measured with an electronic force sensing probe(Yeaple Probe):10, 20, 30, 40,up to 50 grams of force are applied to hypersensitive tooth until pain is felt. This calibrated instrument measures grams of force applied to each tooth before pain is felt. This data is recorded as the hypersensitivity score. The lower the score, the higher the hypersensitivity.Changes in this score to potentially painful stimulus are determined based on how many grams of force can be applied before the subject reports feeling pain. Grams of force is therefore the unit measurement for sensitivity
Time Frame: 12 weeks (Final)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nupro C Prophylaxis Paste | ProClude Prophylaxis Paste
Number analyzed (Participants) | 35 | 44
Units on a scale | 10.83 (1.89) | 10.63 (2.11)
Statistical Analysis 1: Comparison: Nupro C Prophylaxis Paste vs ProClude Prophylaxis Paste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

2. Primary Outcome: Tooth Hypersensivity Stimuli to Air
Description: Units on a scale using Schiff Cold Air Sensitivity Scale. Response to a constant (duration, pressure, temperature, distance from target) jet of air applied to a hypersensitive tooth. According to this analog scale hypersensitivity scores for the stimulated tooth is 0, 1, 2 or 3(The lower the score, the lower the hypersensitivity). 0=No subject response to stimulus, 1=responds but will continue, 2=responds and moves or requests discontinuation, 3=Painful response to stimulus, discontinuation requested.
Time Frame: 12 weeks (Final)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nupro C Prophylaxis Paste | ProClude Prophylaxis Paste
Number analyzed (Participants) | 35 | 44
Units on a scale | 2.69 (0.32) | 2.73 (0.36)
Statistical Analysis 1: Comparison: Nupro C Prophylaxis Paste vs ProClude Prophylaxis Paste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Nupro C Prophylaxis Paste | ProClude Prophylaxis Paste
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/44
Other Adverse Events (participants affected / at risk) | 0/35 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days